CLINICAL TRIAL: NCT06660342
Title: Vonoprazan Pregnancy Registry: An Observational Study of the Safety of Vonoprazan Exposure in Pregnant Women and Their Offspring
Brief Title: A Study of the Safety of Vonoprazan Exposure in Pregnant Women and Their Offspring
Status: Recruiting | Type: Observational
Sponsor: Phathom Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VONO-402
Record Dates: First submitted 2024-10-22; First posted 2024-10-28 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Erosive Esophagitis; Heartburn; Symptomatic Non-erosive Gastroesophageal Reflux Disease; Helicobacter Pylori Infection
Keywords: Erosive Esophagitis; Heartburn; Symptomatic Non-erosive Gastroesophageal Reflux Disease; Helicobacter Pylori Infection; Pregnant Women; Fetal; Infant
MeSH Terms: conditions — Heartburn | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed Cohort: Pregnant women who are exposed to vonoprazan during pregnancy.
  Interventions: Drug: Vonoprazan
- Unexposed Cohort: Pregnant women who are not exposed to vonoprazan during pregnancy but who may be exposed to other products for the treatment of conditions for which vonoprazan may be prescribed.

INTERVENTIONS:
Drug: Vonoprazan — Oral tablet.
  Groups: Exposed Cohort

SUMMARY:
The main objective of the study is to compare the maternal, fetal, and infant outcomes of pregnant women who are exposed to vonoprazan during pregnancy with outcomes of an internal comparison cohort of pregnant women who are unexposed to vonoprazan during pregnancy but who may be exposed to other products for the treatment of conditions for which vonoprazan may be prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Women 15 to 50 years of age.
* Currently or recently pregnant.
* Consent to participate.
* Authorization for her health care provider(s) (HCP[s]) to provide data to the registry.
* Exposed cohort: Exposure to at least one dose of vonoprazan during pregnancy.
* Unexposed cohort: Unexposed to vonoprazan and diagnosis of any condition for which vonoprazan may be prescribed.

Exclusion Criteria:

* Occurrence of pregnancy outcome prior to first contact with the virtual research coordination center (VRCC) (retrospectively enrolled).
* Exposure to known tetratogens and/or investigational medications during pregnancy.
* Lost to follow-up.

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study aims to enroll a total of 728 pregnant women in the study population from the United States, with 364 women in each cohort. This sample size will afford the study the ability to detect a 3-fold increase in the prevalence of the primary outcome, MCM, in the exposed cohort with 80% power.
Sampling Method: Non-Probability Sample
Enrollment: 728 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2034-09 (Estimated); Study Completion 2034-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Major Congenital Malformations (MCMs) | Date of conception (DOC) to pregnancy outcome for fetal losses (approximately 40 gestational weeks) or 12 months from birth for live births

SECONDARY OUTCOMES:
Number of Participants with Minor Congenital Malformations | DOC to pregnancy outcome for fetal losses (approximately 40 gestational weeks) or 12 months from birth for live births
Number of Participants who Experience Spontaneous Abortion (SAB) | DOC to 19 gestational weeks
Number of Participants who Experience Stillbirth | 20 gestational weeks to pregnancy outcome (approximately 40 weeks)
Number of Participants who Experience Elective Termination | DOC to pregnancy outcome (approximately 40 weeks)
Number of Participants who Experience Preterm Birth | DOC to 36 gestational weeks
Number of Participants who are Small for Gestational Age (SGA) | At delivery of live birth (approximately 40 weeks)
Number of Participants who Experience Postnatal Growth Deficiency | 4 Months and 12 Months from Birth
Number of Participants who Experience Infant Developmental Delay | 4 Months and 12 Months from Birth

CONTACTS AND LOCATIONS:
Locations (1):
- PPD, Wilmington, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No